CLINICAL TRIAL: NCT01677806
Title: Investigational Percutaneous Vertebroplasty Efficacy and Safety Trial
Brief Title: Safety and Efficacy Study of Percutaneous Vertebroplasty for Painful Acute Osteoporotic Spine Fractures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jinan Military General Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); Shanghai 10th People's Hospital (Other); China Medical University, China (Other); Beijing Friendship Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Gang Sun;Chungen Wu;Maoquan Li;Bo Feng; Hai Tang;ZL Deng, Clinical Professor, Jinan Military General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JNMGH20120821
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Acute Osteoporotic Spinal Fractures
Keywords: Percutaneous vertebroplasty
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous vertebroplasty (Experimental)
  Interventions: Procedure: Percutaneous vertebroplasty
- Conservative therapy (Active Comparator)
  Interventions: Other: Conservative therapy

INTERVENTIONS:
Procedure: Percutaneous vertebroplasty — Percutaneous vertebroplasty Placement of PMMA into vertebral compression fracture
  Arms: Percutaneous vertebroplasty
Other: Conservative therapy — Conservative therapy mainly consists of optimal pain medication. Pain management is titrated according to patients' needs, including analgesia, bed rest, and physical support (bracing).
  Arms: Conservative therapy

SUMMARY:
Percutaneous vertebroplasty (PVP) is now a therapeutic option for individuals for whom medical management has not been successful or for those who are at risk for developing complications due to long-term immobilization. Recently, three randomized controlled trials (RCT) concerning PVP have been published with conflicting results. Two RCTs with a sham control intervention failed to show an advantage of vertebroplasty over placebo for participants with acute, subacute, and chronic fractures or severe pain. In the third RCT, PVP compared to optimal conservative treatment showed significant immediate postoperative pain relief in the vertebroplasty group, but not at 3 and 12 months. To examine these issues, this study is initiated to compare PVP with conservative therapy in patients with osteoporotic VCFs. Moreover, this study addresses concerns about the possibility that PVP increases the incidence of new compression fractures in adjacent vertebrae.

DETAILED DESCRIPTION:
Osteoporotic vertebral fractures (OVCFs) are common in the elderly population, with an estimated 1.4 million new fractures occurring every year worldwide. Patients may present with pain and frequently require hospital admission for analgesia, bed rest, and physical support (bracing). While their back pain may last for 6-12 weeks, complications such as pneumonia, decubitus ulcers, venous thromboembolism, and even death may occur. Percutaneous vertebroplasty (PVP) is now a therapeutic option for individuals for whom medical management has not been successful or for those who are at risk for developing complications due to long-term immobilization. Recently, three randomized controlled trials (RCT) concerning PVP have been published with conflicting results. So this study is to compare PVP with conservative therapy in patients with osteoporotic VCFs. Moreover, this study addresses concerns about the possibility that PVP increases the incidence of new compression fractures in adjacent vertebrae.

This study is a multicenter randomized controlled trial (RCT), Participants in this study will be allocated randomly to PVP or conservative treatment.All Participants will be asked to fill out standard questionnaires to provide clinical information at baseline (the day of randomization), and at 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after the treatment. Cross-over will not be offered before 12 months after randomization. All standard questionnaires (except the 1-day questionnaire) consist of the VAS score, Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO), EQ-5D, and Roland-Morris Disability (RMD) Questionnaire. Furthermore,additional questions about pain treatment, hospital stay, outpatient visits,medical aids, and medical costs will be completed with the help of a nurse practitioner.

ELIGIBILITY:
Inclusion Criteria:

* 50 Years and older
* have a confirmed diagnosis of osteoporosis or osteopenia.
* acute, painful OVCFs from T4-L5
* clinical onset < 6 weeks
* vertebral compression fracture on spine radiograph (minimum 15% height loss)
* Visual Analogue Scale [VAS] score ≥ 4 for pain

Exclusion Criteria:

* severe cardio-pulmonary condition
* untreatable coagulopathy
* active local or systemic infection
* current malignancy, or radicular or caudal compression syndrome

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
VAS score | at 1 month
  Pain assessment is based on the VAS scale, a scale from 0 (no pain) to 10 (worst pain ever), for which a decrease of 3.0 or more points from baseline is considered to be clinically significant pain relief.

SECONDARY OUTCOMES:
QUALEFFO total score | at baseline, 1 week, 1 month, 3 months, 6 months, and 12 months after the treatment.
  QUALEFFO total score is measured with the Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO). This questionnaire consists of 41 items and includes five domains: pain, physical function, social function, general health perception, and mental function.
ED-5Q score | at baseline, 1-week, and 1-, 3-, 6-, and 12- month
  EQ-5D is a standardized instrument utilized as a measure of health-related quality of life outcomes. Furthermore, EQ-5D is one of a few measures recommended for use in cost-effectiveness analyses by the Washington Panel on Cost Effectiveness in Health & Medicine as well as in National guidelines in economic evaluation.
RMD score | at baseline, 1-week, and 1-, 3-, 6-, and 12- month
  The RMD questionnaire is a disability questionnaire that measures the functional status of patients with back pain. RMD scores range from 0 to 24, with higher numbers indicating worse physical functioning.
New vertebral fractures | at baseline, 1 month, 3 months, and 1 year.
  New vertebral fractures are defined as a decrease (compared with baseline radiographs) of 20% or more, and at least 4 mm, in any of the three vertebral heights (anterior, middle, or posterior) on follow-up.
Total medical costs | at 1-month, 12-month
  This study will calculate total medical costs through summarizing all costs of drugs,family doctor,physiotherapist, hospital stay, and outpatient visits, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Sun, M.D, Principal Investigator — The Jinan Military General Hospital
Locations (1):
- The Jinan Military General Hospital, Jinan, Shandong, China